CLINICAL TRIAL: NCT07216950
Title: Knowledge and Interpersonal Skills to Develop Enhanced Relationships (KINDER): Testing the Efficacy of an Intervention to Prevent Psychological Elder Abuse in Family Caregiving
Brief Title: Knowledge and Interpersonal Skills to Develop Enhanced Relationships (KINDER)
Acronym: KINDER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kylie Meyer, Principal Investigator, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY20250080
Record Dates: First submitted 2025-10-12; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Elder Mistreatment; Elder Abuse; Quality of Care; Dementia; Caregiving
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KINDER Intervention Arm (Experimental): KINDER is an 8-week intervention that consists of three facilitated group discussion sessions conducted over Zoom with a small group of caregivers, in addition to self-paced lessons delivered using a printed or PDF workbook, depending on participant preference. Throughout KINDER, caregivers reflect on their relationship, including how their behavior toward the care recipient may need to change considering new vulnerabilities with dementia, and how to communicate about topics that often contribute to conflict, such as balancing safety and independence (e.g., driving).
  Interventions: Behavioral: Knowledge and Interpersonal Skills to Develop Enhanced Relationships
- Control Condition (Placebo Comparator): Caregivers in the control arm will receive a workbook that covers 8 weeks of content focused on healthy living (e.g., nutrition).
  Interventions: Behavioral: Healthy Living for the Caregiver

INTERVENTIONS:
Behavioral: Knowledge and Interpersonal Skills to Develop Enhanced Relationships — KINDER is an 8-week intervention that consists of three facilitated group discussion sessions conducted over Zoom with a small group of caregivers, in addition to self-paced lessons delivered using a printed or PDF workbook, depending on participant preference. Throughout KINDER, caregivers reflect on their relationship, including how their behavior toward the care recipient may need to change considering new vulnerabilities with dementia, and how to communicate about topics that often contribute to conflict, such as balancing safety and independence (e.g., driving).
  Arms: KINDER Intervention Arm
Behavioral: Healthy Living for the Caregiver — Caregivers in the control arm will receive a workbook that covers 8 weeks of content focused on healthy living (e.g., nutrition).
  Arms: Control Condition

SUMMARY:
The Knowledge and Interpersonal Skills to Develop Enhanced Relationships (KINDER) intervention was developed to prevent psychological elder abuse (EA) and promote high-quality caregiving by lowering relationship strain and developing CG resourcefulness. The goal of this two-arm, randomized control trial is to determine the efficacy of KINDER at mitigating psychological EA by family caregivers to persons living with dementia and to describe how the intervention may work to reduce psychological EA.

ELIGIBILITY:
Inclusion Criteria:

* Family member, including family of choice, to an individual living with AD/ADRD
* Is aged 18 years or older;
* Provides assistance with at least two instrumental activities of daily living or one activity of daily living;
* Provides at least 4 hours of caregiving per day
* The care recipient is at least age 65 or older
* The care recipient has early or mid-stage AD/ADRD, as indicated by a score of 4 to 6 on the Global Deterioration Scale

Exclusion Criteria:

* Sees the care recipient in-person less than 2 times per week
* Has plans to place the care recipient in a skilled nursing facility within the next 8 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2026-03-11 (Estimated); Primary Completion 2028-11-11 (Estimated); Study Completion 2029-05-11 (Estimated)

PRIMARY OUTCOMES:
Psychological Elder Abuse | Baseline, 2 weeks post-intervention, 12 weeks post-intervention, 24 weeks post-intervention
  The investigators will use a modified version of the Conflict Tactics Scale 2 to measure psychological EA (MCTS 2). This scale includes five psychological EA behaviors, such as insulting, swearing at, or yelling at the care recipient, as well as threatening to stop taking care of the care recipient, placing them in a nursing home, threatening physical harm, and stomping out of the room. Participants will be asked to describe the frequency of each behavior in the last 2 months, such that response options will include: None, Once, Twice, 3 to 5 times, 6 to 10 times, and More than 10 times. Scores range from 0 to 30. Higher scores indicate greater frequency of mistreatment. Higher scores indicate greater frequency of abuse. The outcome measure will use the average change score from baseline scores until each post-intervention survey.
Quality of Caregiving | Baseline, 2 weeks post-intervention, 12 weeks post-intervention, 24 weeks post-intervention
  To measure quality of care, the investigators will use the 11-item Exemplary Caregiving Scale, which focuses on providing care that meets the care recipient's needs (α=0.73) and is respectful (α=0.76). Response options include Never, Sometimes, Often, and Always (range: 11 to 44). Higher scores indicate higher quality of caregiving. The outcome measure will use the average change score from baseline scores until each post-intervention survey.

SECONDARY OUTCOMES:
Resourcefulness | Baseline, 2 weeks post-intervention, 12 weeks post-intervention, 24 weeks post-intervention
  Resourcefulness is measured using the 28-item Caregiver Resourcefulness Scale (α=0.85). This scale has two factors: one focused on help-seeking and another on self-help. Caregivers are asked the frequency at which they use different strategies to manage challenges, and may respond: Not at all like me (0), Pretty much not like me (1), A little bit not like me (2), A little bit like me (3), Pretty much like much like me (4), or Very much like me (5). Items are added together to create a total score. Scores range from 0 to 140, where higher scores indicate higher levels of resourcefulness. The outcome measure will use the average change score from baseline scores until each post-intervention survey.
Caregiving Relationship Strain | Baseline, 2 weeks post-intervention, 12 weeks post-intervention, 24 weeks post-intervention
  Relationship strain will be measured using the 5-item Strain Scale of the Dyadic Relationship Scale (α=0.69). Respondents are asked to indicate agreement with statements such as, "The patient made too many requests," and may indicate Strongly Disagree, Disagree, Agree, or Strongly Agree. The scale has a range of scores from 4 to 20, where higher scores indicate greater levels of relationship strain. The outcome measure will use the average change score from baseline scores until each post-intervention survey.

OTHER OUTCOMES:
Other Types of Elder Abuse | Baseline, 2 weeks post-intervention, 12 weeks post-intervention, 24 weeks post-intervention
  Other types of elder abuse will be measured with the Geriatric Mistreatment Scale (GMS). The GMS is a 22-items scale that measures psychological, physical, sexual, financial abuse, and neglect using "yes" and "no" questions (range of response: 0 to 22). Higher scores indicate greater frequency of abuse. The outcome measure will use the average change score from baseline scores until each post-intervention survey.
Depressive Cognitions | Baseline, 2 weeks post-intervention, 12 weeks post-intervention, 24 weeks post-intervention
  Caregiver depressive cognitions will be measured using the Depressive Cognitions Scale, which measures thinking patterns preceding depression. The 8-item Depressive Cognitions Scale is validated for use among AD/ADRD CGs, with a Cronbach's alpha of 0.75 to 0.88. Respondents indicate their level of agreement with each statement on a 6-point Likert scale with responses from "totally disagree" to "totally agree." Scores range from 0 to 40. Higher scores indicate higher levels of depressive cognitions. The outcome measure will use the average change score from baseline scores until each post-intervention survey.
Social Support | Baseline, 2 weeks post-intervention, 12 weeks post-intervention, 24 weeks post-intervention
  Social Support will be measured using the NIH Toolbox measure for emotional support. This scale has 8 items about how frequently individuals access support (e.g., someone who understands my problems). Scores range from Never, Rarely, Sometimes, Usually, and Always (range=8-40). Higher scores indicate higher levels of social support. The outcome measure will use the average change score from baseline scores until each post-intervention survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Baseline and follow up surveys with participants; Referral, screening, enrollment, and retention data; Fidelity surveys. All data will be de-identified.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Information will be shared no later than the time of an associated publication or the end of the performance period, whichever comes first. Data will be made available indefinitely.
Access Criteria: Survey data and metadata will be shared through National Archive of Computerized Data on Aging (NACDA) as open access. Once prepared, data will be released by NACDA. NACDA users must register and agree to the Terms of Use, such as agreeing not to attempt to identify individual participants. Data users also agree not to share or redistribute data downloads